CLINICAL TRIAL: NCT00846547
Title: An Open-Label, Flexible-Dose Evaluation of the Safety and Tolerability of STX209 for Treatment of Irritability in Subjects With Autism Spectrum Disorders
Brief Title: Open-Label Study of the Safety and Tolerability of STX209 in Subjects With Autism Spectrum Disorders
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Seaside Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22003
Record Dates: First submitted 2009-02-17; First posted 2009-02-18 (Estimated); Results first posted 2013-06-14 (Estimated); Last update posted 2013-06-14 (Estimated); Status verified 2013-05

CONDITIONS: Autism Spectrum Disorders
Keywords: Autism; Autism Spectrum Disorders; irritability; aberrant behavior
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder | interventions — arbaclofen placarbil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arbaclofen (Experimental)
  Interventions: Drug: Arbaclofen

INTERVENTIONS:
Drug: Arbaclofen — variable dose from 1mg bid to 10 mg tid, oral capsule, 8 week treatment period
  Other Names: STX209

SUMMARY:
The study objective is to explore the safety and tolerability of STX209 in subjects with Autism Spectrum Disorders and to obtain preliminary data on several measures of efficacy in treating irritability. We hypothesize that STX209 will be safe and well-tolerated.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects 6 to 17 years of age, inclusive.
* Diagnosis of Autistic spectrum disorders
* Clinical Global Impression - Severity (CGI-S) rating for aberrant behavior of moderate or higher at screening and at Visit 1 (Day 1).
* An Aberrant Behavior Checklist (ABC-C) Irritability Subscale score ≥16 at screening and at Visit 1 (Day 1).
* If the subject is already receiving stable non-pharmacologic educational, behavioral, and/or dietary interventions, participation in these programs must have been continuous during the 3 months prior to Screening (Visit 1) and subjects and their parent/caregiver/legally authorized representative (LAR) will not electively initiate new or modify ongoing interventions for the duration of the study.
* Exclusion Criteria:
* Subjects with known genetic disorders associated with PDD such as fragile X syndrome.
* Subjects with a history of a seizure disorder who are not currently receiving treatment with antiepileptic medication.
* Subjects with any medical condition, including alcohol and drug abuse that might interfere with the conduct of the study, confound interpretation of the study results, or endanger their own well-being.
* Subjects who plan to initiate or change pharmacologic or non-pharmacologic interventions during the course of the study.
* Subjects currently treated or have been treated in the last 2 weeks with any psychotropic medication except anti-epileptics or who have been treated with fluoxetine in the last 4 weeks.
* Subjects currently treated with vigabatrin or tiagabine.
* Subjects taking another investigational drug currently or within the last 30 days.
* Subjects who have a history of hypersensitivity to racemic baclofen.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 32 (Actual)
Dates: Start 2009-02; Primary Completion 2010-06 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence Scahill, PhD, Principal Investigator — Yale University; Craig Erikson, MD, Principal Investigator — Riley Hospital for Children; Bryan King, MD, PhD, Principal Investigator — Seattle Children's Hospital; James McCracken, MD, Principal Investigator — University of California, Los Angeles; Linmarie Sikich, MD, Principal Investigator — University of North Carolina Neurosciences Hospital; Jeremy Veenstra-VanderWeele, MD, Principal Investigator — Vanderbilt Kennedy Center; Lawrence Ginsberg, MD, Principal Investigator — Red Oaks Psychiatry Associates, PA; Raun Melmed, MD, Principal Investigator — Southwest Autism Research & Resource Center
Locations (8):
- United States (8):
  - Southwest Autism Research & Resource Center, Phoenix, Arizona
  - University of California-Los Angeles Neuropsychiatric Institute, Los Angeles, California
  - Yale Child Study Center, New Haven, Connecticut
  - Riley Hospital for Children, Indianapolis, Indiana
  - University of North Carolina Neurosciences Hospital, Chapel Hill, North Carolina
  - Vanderbilt Kennedy Center, Nashville, Tennessee
  - Red Oaks Psychiatry Associates, PA, Houston, Texas
  - Seattle Children's Hospital, Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Groups:
- Arbaclofen: Arbaclofen (STX209) : variable dose from 1mg bid to 10 mg tid, oral capsule, 8 week treatment period
Period: Overall Study
Arm/Group | Arbaclofen
Started | 32
Completed | 25
Not Completed | 7

BASELINE CHARACTERISTICS:
Arm/Group | Arbaclofen
Number analyzed (Participants) | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 32
  Between 18 and 65 years | 0
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 11.8 (3.13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 29
Region of Enrollment [Number; unit: participants]
  United States | 32

OUTCOME MEASURES:

1. Primary Outcome: Irritability Subscale of the Aberrant Behavior Checklist, Community Version
Description: The Aberrant Behavior Checklist-Community Edition (ABC-C) is a 58-item questionnaire composed of five different independent subscales. The questionnaire is completed by the parent/caregiver and lists aberrant behaviors and asks about the severity of the problem. ABC-Irritability is one of the subscales and comprises of 15 items. Minimum score is 0, maximum is 45. A decreased score indicates few aberrant behaviors and clinical improvement. The entire ABC-C assessment is administered at baseline and then at the end of each Intervention Period (4 weeks after Baseline).
Time Frame: At 8 weeks during the treatment period
Measure: Least Squares Mean (Standard Error); unit: Points on a scale
Arm/Group | Arbaclofen
Number analyzed (Participants) | 32
Points on a scale | -8.9 (1.73)

ADVERSE EVENTS:
Arm/Group | Arbaclofen
Serious Adverse Events (participants affected / at risk) | 1/32
Other Adverse Events (participants affected / at risk) | 28/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arbaclofen (N=32)
increased aggression (Psychiatric disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arbaclofen (N=32)
agitation (Psychiatric disorders) | 7
irritability (Psychiatric disorders) | 7
psychomotor hyperactivity (Psychiatric disorders) | 5
insomnia (Psychiatric disorders) | 4
aggression (Psychiatric disorders) | 3
disturbance in attention (Psychiatric disorders) | 3
self injurious behaviour (Psychiatric disorders) | 2
diarrhoea (Gastrointestinal disorders) | 4
abdominal pain upper (Gastrointestinal disorders) | 2
vomiting (Gastrointestinal disorders) | 2
nasopharyngitis (Infections and infestations) | 3
pharyngitis streptococcal (Infections and infestations) | 2
upper respiratory tract infection (Infections and infestations) | 2
fatigue (General disorders) | 5
headache (Nervous system disorders) | 3
dizziness (Nervous system disorders) | 2
cough (Respiratory, thoracic and mediastinal disorders) | 2
decreased appetite (Metabolism and nutrition disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Seaside Therapeutics agreements with investigators vary; constant is our right to restrict communications regarding trial results prior to public release for ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.